CLINICAL TRIAL: NCT05791630
Title: The Norwegian World Health Organisation Labour Care Guide Trial
Brief Title: The Norwegian World Health Organisation Labour Care Guide Trial (NORWEL)
Acronym: NORWEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Stine Bernitz, Professor/researcher, Ostfold Hospital Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023084
Record Dates: First submitted 2023-01-17; First posted 2023-03-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Labor Dystocia; Labor Complication; Labor Onset and Length Abnormalities; Labor (Obstetrics)--Complications; Experience, Life; Progression; Cesarean Section Complications; Apgar; 4-7 at 1 Minute
MeSH Terms: conditions — Dystocia; Obstetric Labor Complications; Disease Progression

STUDY DESIGN:
Intervention Model Description: Multicenter stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WHO partograph (No Intervention): all study sites use the WHO partograph as standard care in the first step of the trial
- WHO labour care guide (Experimental): All study sites will cross over to the intervention according to randomization and use the LCG for assessing labour progression and wellbeing in labour
  Interventions: Other: the labour care guide (LCG)

INTERVENTIONS:
Other: the labour care guide (LCG) — The labour care guide is a tool to be used for assessing labour progression and monitoring care in labour
  Arms: WHO labour care guide

SUMMARY:
Appropriate and timely care during birth is critical to the survival and health of women and their babies. In 2020, the World Health Organization (WHO) presented the Labour Care Guide (LCG) as the new recommended tool for monitoring birth and assessing progression, replacing the WHO partograph. This evidence-based guide was designed to ensure improved quality and safety of care, and to avoid unnecessary interventions during birth. The LCG was developed to be used in all settings globally, but it has only been tested in health facilities in South America, Asia and Africa, while it has not been tested in high-income settings. Implementing a new guideline for monitoring birth is a comprehensive operation that will affect both the national economy, health systems, and individual patients; therefore, further research on the possible advantages is needed before national enrolment. Hence, the trial proposed in this application is crucial to form the required foundation of knowledge. The trial will be conducted in labour wards at ten hospitals, covering all health regions in Norway, and the established Norwegian Research Network for Clinical Studies in Obstetrics (NORBIRTH), with dedicated local principal investigators, will provide a robust research environment. This trial will test the effect of the LCG. Results from this trial will provide knowledge needed to determine a future implementation of the LCG in Norway.

DETAILED DESCRIPTION:
A large robust trial investigating the effect of the LCG is needed to establish a foundation of knowledge on which the decision of implementing the LCG on a national level should be based. The Norwegian WHO LCG trial addresses the WHO research priority question: "What is the effect of the LCG on processes of care, health, well-being and outcomes during labour and childbirth?". The trial will have a special focus on intrapartum caesarean section rates and experience of labour.

The overall aim of the trial is to test the LCG in an unbiased population in a Norwegian setting. The project will conduct a nationwide randomized controlled trial (RCT) to test the effect on labour interventions and maternal and neonatal outcomes compared to the previous WHO partograph. The Norwegian WHO LCG trial will be conducted through three work packages: WP1 consists of a feasibility study to develop an electronic version of the LCG, and will test its validity and usability prior to the planned RCT. WP2 consists of a stepped wedge RCT to assess the effect of the LCG on labour interventions and maternal and neonatal outcomes. WP3 consists of a survey to investigate patient reported outcome through the childbirth experience questionnaire (CEQ).

This is a stepped wedge multicenter cluster randomised non-inferiority trial, to be conducted within the nationwide NORBIRTH network for clinical obstetric research. The hospitals will act as clusters and the women as individual participants.

During the trial period all hospitals will use the WHO partograph and the LCG according to the trial protocol for all women with a planned vaginal delivery, these women constitute the trial population. Women who want to opt out will not be included in the analyses. Each hospital has established local research groups which are dedicated to implement the project. The included hospitals will consent to adhere to the protocol in the trial period and state that they have the capacity to participate both logistically and practically. Local coordinators will be appointed with the responsibility of monitoring the trial and secure a thorough documentation according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women in active labour
* Labour and delivery at study sites

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women in labour and delivery
Enrollment: 23650 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Intrapartum cesarean section | 18 months
  the rate of intrapartum cesarean sections (ICS), presented in numbers and percentages.

SECONDARY OUTCOMES:
Instrumental vaginal delivery | 18 months
  The rate of instrumental vaginal delivery, presented in numbers and percentages
Perineal tears | 18 months
  Perineal tears will be presented in numbers and percentages
Post partum hemorrhage | 18 months
  Post partum hemorrhage will be presented in numbers and percentages.
Estimated blood loss | 18 months
  Estimated blood loss will be presented in ml of blood loss
Blood transfusion | 18 months
  The need for blood transfusion will be presented in numbers and percentages
The use of oxytocin | 18 months
  The use of oxytocin will be presented in numbers and percentages
Dosage of oxytocin | 18 months
  The dosages of oxytocin will be presented in milli units (m/U)
Duration of oxytocin | 18 months
  The duration of oxytocin will be presented in hours and minutes
initiation of oxytocin | 18 months
  Initiation of oxytocin will be presented according to cervical dilatation in centimetres
Labour duration | 18 months
  Labour duration will be presented in hours and minutes
The use of epidural analgesia | 18 months
  The use of epidural analgesia will be presented in numbers and percentages
Duration of epidural analgesia | 18 months
  Duration of epidural analgesia will be presented hours and minutes
Initiation of epidural analgesia | 18 months
  The initiation of epidural analgesia will be presented according to cervical dilatation presented in centimetres
The use of medical pain relief in labour | 18 months
  The use of medical pain relief will be presented in numbers and percentages.
The use of non-medical pain relief in labour | 18 months
  The use of non-medical pain relief will be presented in numbers and percentages.
Childbirth experience | 20 months
  Childbirth experience measured by the childbirth experience questionnaire, CEQ presented in total and mean scores according to the four domains in the CEQ questionnaire
Intermittent fetal monitoring | 18 months
  The use of intermittent fetal monitoring (pinard and doppler) will be presented in numbers and percentages
Continuous fetal monitoring | 18 months
  The use of continuous fetal monitoring will be presented in numbers and percentages
Neonatal Apgar scores | 18 months
  Apgar scores 1/5/10 minutes post partum presented in values of 0-10
Neonatal metabolic acidosis | 18 months
  Metabolic acidosis will be presented in numbers and percentages
Admittance to Neonatal Intensive Care Unit | 18 months
  Admittance to the Neonatal Intensive Care Unit will be presented in numbers and percentages
Duration of stay at neonatal Intensive Care Unit | 18 months
  Duration of stay at neonatal Intensive Care Unit will be presented days
Neonatal gender | 18 months
  Neonatal gender will be presented by numbers and percentages
Neonatal birth weight | 18 months
  Neonatal birth weight will be presented in kilograms
Neonatal birth head circumference | 18 months
  Neonatal head circumference will be presented in centimetres
Neonatal morbidity | 18 months
  Neonatal morbidity will be presented in numbers and percentages.

OTHER OUTCOMES:
Continuous support in labour | 18 months
  Continuous support will be presented as yes/no and according to cervical dilatation
Birthing position | 18 months
  The birthing position will registered and presented in numbers and percentages
Fetal presentation | 18 months
  The fetal delivery presentation will be registered and presented in numbers and percentages
Perineal support | 18 months
  Perineal support will be registered in numbers and percentages
Skin-to-skin-contact | 18 months
  Immediate skin-to-skin-contact will be registered as yes/no and time for immediate skin-to-skin-contact will be presented in hours and minutes
Breast feeding | 18 months
  Breastfeeding will be presented as number and percentages
The use of formula | 18 months
  The use of formula will be registered as number and percentages
Usability of the Labour Care Guide | 24 months
  Midwives' and doctors' experience with LCG use assessed through a customized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stine Bernitz, PhD, Principal Investigator — Ostfold Hospital Trust
Locations (10):
- Norway (10):
  - Akershus University Hospital, Ahus, Nordbyhagen, Akershus
  - Vestre Viken Helseforetak, Drammen, Drammen, Buskerud
  - Sørlandet Hospital Kristiansand, Kristiansand, Kristiansand
  - Oslo university hospital Rikshospitalet, Oslo, Oslo County
  - Oslo University Hospital Ullevål, Oslo, Oslo County
  - Stavanger University Hospital, Stavanger, Rogaland
  - University Hospital Northern Norway, Tromsø, Tromsø, Troms
  - St.Olav University Hospital, Trondheim, Trøndelag
  - Haukeland University Hospital, Bergen, Vestland
  - Ostfold Hospital Trust, Greåker, Østfold fylke

IPD SHARING:
Plan to Share IPD: Yes
Will be shared according to demand and aim
Supporting Information: Study Protocol, ICF, CSR
Time Frame: from onset of trial until five years after the trial has ended
Access Criteria: if the purpose is stated and acceptable and presented by scientific personnel